CLINICAL TRIAL: NCT06902649
Title: Step-by-Step: Evaluation of a Stepped Care Model for Anger, Defiant, or Aggressive Behavior in Children and Adolescents
Brief Title: Step-by-Step: Evaluation of a Stepped Care Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Pia Enebrink, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00381-01
Record Dates: First submitted 2025-03-21; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Child Behavior Problem; Disruptive Behavior; Oppositional Defiant Disorder; Conduct Problems; Aggression; Anger
Keywords: Disruptive Behavior; Child Behavior Problem; Cognitive behavior therapy; Virtual Reality; Parenting support program
MeSH Terms: conditions — Problem Behavior; Oppositional Defiant Disorder; Aggression | interventions — Methods; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Internet-based parenting support (Experimental): 5 weeks of internet-based parenting support provided as a first step for all parents (Step 1 in the stepped care model).
  Interventions: Behavioral: Internet-based parenting support
- "YourSkills" for children/youth (Experimental): A cognitive-behavioral program for children and youth with up to 10 individual, face-to-face, weekly sessions, where role-plays can be conducted in virtual reality. (Step 2 in the stepped care model)
  Interventions: Behavioral: "YourSkills" for children/youth
- Step-by-step parent support (Experimental): A parent training program with between 6 and 10 individual, face-to-face, weekly sessions with parents. Role-plays may be conducted in virtual reality. (Step 2 in the stepped care model)
  Interventions: Behavioral: Step-by-step parent support
- Intervention/supports as usual and prolonged use of internet-based parenting support (Active Comparator): Based on other available support at the units and prolonged use of internet-based parenting support program. (Step 2 in the stepped-care model)
  Interventions: Behavioral: Intervention/support as usual and prolonged use of internet-based parenting support

INTERVENTIONS:
Behavioral: Internet-based parenting support — An internet-based parent training program with 5 active modules and a final summarizing module, based on social learning theory/cognitive behavior therapy. All parents participate in this intervention (Step 1) before being randomized to the other three arms of the stepped care model in the randomized controlled trial (Step 2).
  Arms: Internet-based parenting support
Behavioral: "YourSkills" for children/youth — Cognitive behavioral therapy for children/youth with role-plays in virtual reality. A program for children/youth with anger problems or aggressive behaviors based on social learning theory and cognitive behavior therapy (CBT), incorporating virtual reality (VR) when conducting brief role-plays. The program includes similar strategies as other CBT-oriented programs for anger problems, with the addition of VR for practicing skills.
  Arms: "YourSkills" for children/youth
Behavioral: Step-by-step parent support — A parent training program based on social learning theory and cognitive behavioral therapy (CBT), including some sessions where virtual reality may be used for training in brief role plays. The program includes similar strategies as other common CBT-parent training programs for parents of children with behavior problems, with the difference that virtual reality can be used as an additional way to practice skills.
  Arms: Step-by-step parent support
Behavioral: Intervention/support as usual and prolonged use of internet-based parenting support — Based on other available support, interventions, courses at the units. Parents have access to the internet-based parenting support provided in Step 1 (the first intervention of the study). After 10 weeks with intervention/support as usual, the parents are asked if they want to participate in the CBT-VR-intervention for children (YourSkills) or for parents (Step-by-Step parent support).
  Arms: Intervention/supports as usual and prolonged use of internet-based parenting support

SUMMARY:
The primary aim of this project is to examine the effectiveness of a stepped care model of interventions for children's defiant or aggressive behavior problems. The stepped model consists of a brief internet-based parenting support program (Step 1). For those with continued need of additional interventions, Step 2 includes access to one of following interventions: b) a Cognitive Behavior Therapy (CBT) -Virtual Reality (VR)-assisted parenting support program, b) a Cognitive Behavior Therapy -Virtual Reality-assisted child intervention, or c) standard interventions/support at the family's unit/clinic and continued access to the study's internet-based parenting support program, after which the family may choose CBT-VR for the child or the parent.

DETAILED DESCRIPTION:
Children who exhibit severe aggressive and defiant behavior from an early age are at increased risk of persistent behavioral problems during adolescence and into young adulthood. Additionally, they are more likely to experience difficulties in social contexts, lack prosocial friendships, fall behind academically in school, and have poorer mental well-being.

Parenting support programs are recommended for parents of children under the age of 12 with oppositional defiant disorder or conduct disorder, as well as for parents of adolescents with less severe behavioral problems. Therefore, such programs can serve as a foundation for interventions offered to parents of children with behavioral problems. However, many parenting support programs are delivered in a group format, are not possible to attend for all parents, have challenges related to parental engagement and dropout, and fewer programs have been evaluated for parents of adolescents.

Cognitive behavioral therapy (CBT) for children with behavioral problems, including anger management training, social skills training, and problem-solving training, have been shown to reduce anger and aggressive behavior and may complement parent support programs for children/youth with behavior problems.

However, there still remains a need for effective stepped care interventions for parents and children/youth with behavior problems.

PURPOSE AND RESEARCH QUESTIONS:

The main aim is to examine the effectiveness of a stepped care model of interventions for families with children/youth aged 8-16 years with behavioral problems, consisting of (Step 1) a brief internet-based parenting support program, and thereafter access to one of following interventions: a) a Cognitive Behavior Therapy (CBT)-Virtual Reality (VR)-assisted parenting support program, b) a CBT-VR-assisted child intervention, or c) standard interventions/support at the family's unit/clinic and continued access to the study's internet-based parenting support program (Step 2). The specific research questions are as follows:

1. What is the effect of the internet-based parenting support program (Step 1), the CBT-VR parenting support program, and the CBT-VR child intervention over time and compared to standard interventions/support (Step 2), on children's behavioral problems, emotional and overall well-being, parental emotion regulation, wellbeing, parenting strategies and family conflicts-both immediately after the interventions and six months after Step 2? How are the interventions perceived by parents and children?
2. To what extent do (a) improved emotion regulation, (b) increased warmth in the family, and (c) a reduction in negative parenting styles contribute to a decrease in children's behavioral problems, i.e., do these variables mediate the outcomes?
3. To what extent do (a) the severity of children's behavioral problems, including diagnoses such as attention deficit hyperactivity disorder, oppositional defiant disorder, and conduct disorder, (b) limited prosocial emotions (so-called callous-unemotional traits), (c) the child's age, gender and (d) parents' initial level of positive parenting style contribute to understanding which families benefit more or less from the interventions, i.e., do these variables moderate or predict the outcomes?
4. To what extent is the stepped care model cost-effective?

METHODS:

This is a project evaluating a two-step intervention care model. The evaluation of each intervention is conducted using a within-group design (repeated measurements before, during, and after each intervention) and, in Step 2, also includes between-group comparisons. Participants are recruited through clinics/units where the interventions are conducted.

Brief written information about the study is available on websites and information channels of the participating units. Families with children of the appropriate age, 8-16 years, and behavioral problems, are informed about the study. After the family/caregivers have reviewed detailed written information and consented to the study (written informed consent), the family is contacted by a clinician/research assistant for a screening interview of inclusion and exclusion criteria. All included parents receive Step 1, the internet-based parent-support. After Step 1, families who wish to continue are randomized to receive either CBT-VR for parents, CBT-VR for children, or standard interventions/support at the family's unit/clinic and continued access to the internet-based parenting support program, whereafter they get access to CBT-VR for children or parents if they want to.

The treatment is evaluated quantitatively by parents and children, using validated assessment scales before, during and after each treatment. Additionally, interviews are conducted with a number of parents and children who have agreed to participate.

POWER CALCULATION:

To identify a moderate treatment effect in Step 2 of the child or parent CBT-VR intervention compared to standard interventions/support (p < .05, power = .80), accounting for a 20% dropout rate, 70 families are needed in the CBT-VR parent, CBT-VR child, and standard intervention groups, i.e., 210 families. Assuming that 33-50% of parents will be in need of the second step, a total of 500-750 parents should be included in the first step, pending a drop-out rate of 20%. Data collection will be completed once 210 families have been included in Step 2.

ANALYSES:

Quantitative data will be visually inspected through graphs, mean values of data, slopes, and variation over time. Differences over time and between groups will be analyzed statistically for both Step 1 and 2-interventions, using methods such as nonparametric tests, General Linear Mixed Modeling (GLMM), paired t-tests, Analysis of variance (ANOVA), Mixed models, Linear regression models. Cohen's d and Reliable Clinical Change will be calculated for all interventions to understand the clinical implications of the results. The primary outcome measure will be compared with results from other parenting support studies, i.e., benchmarking.

Moderator analyses will be conducted through ANOVAs, Linear regression models. Mediation analyses will be conducted using the SPSS (Statistical Package for the Social Sciences) add-on PROCESS macro and bootstrapping, and Linear mixed models.

Qualitative interview-data will be analyzed with thematic analysis.

The health economic evaluation will include two analyses: 1) cost-effectiveness analysis and 2) cost-utility analysis with the outcome measure quality-adjusted life years (QALYs).

ELIGIBILITY:
Inclusion Criteria:

* Families with children aged 8-16 years who have difficulty controlling anger or exhibit defiant or aggressive behavior. The child/adolescent meets 3 of the diagnostic criteria for Oppositional Defiant Disorder or 2 criteria for Conduct Disorder indicating aggressive behavior.
* Medication for the child can remain stable.
* Parents need to be able to read and engage with materials in Swedish

Exclusion Criteria:

* Families with children younger than 8 years old or who have already turned 17, or who do not exhibit defiant or aggressive behaviors according to the first inclusion criterion.
* Children with severe depression, suicidal behavior, bipolar disorder, psychosis, eating disorders, severe autism (level 2 and 3), diagnosed intellectual disability, or ongoing criminal behavior assessed to require interventions other than the study's interventions are excluded.
* Children/adolescents with other ongoing psychological treatments for the same condition or assessed by the clinician in need of other interventions
* Parents and children with epilepsy or migraines

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2025-03-27 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Parent: Mean change from baseline in behavior problems on parent-ratings of the Disruptive Behavior Disorder scale (oppositional defiant disorder subscale). | Pre-, mid- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  The oppositional defiant disorder subscale of the Disruptive Behavior Disorder scale is used for assessing children's behavioral problems. The subscale includes 8 items which are rated on a 4-point scale (0 to 3). The total scale sum ranges from 0 to a total maximum sum of 24 with a higher score indicating more behavior problems.
Parent: Mean change from baseline in oppositional defiant disorder and conduct disorder criteria | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  The number of Oppositional defiant disorder criteria (between 0-8) and Conduct disorder criteria (aggressive symptoms; between 0-5). Total number ranges between 0-13 criteria.
Child/youth: Mean change from baseline in child-ratings of anger on the Anger Expression Scale for children | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program)
  The Anger expression scale for children includes 26 questions about anger and anger management and is rated by children on a 4-point Likert scale (from 1 to 4). Two modified sub-scales are used: anger expression (score ranges from 17 to 68) and anger control (score ranges from 9 to 36) with higher scores indicating higher levels of anger expression and anger control.

SECONDARY OUTCOMES:
Parent: Mean change from baseline in parent-ratings of child wellbeing on the Strengths and Difficulties Questionnaire (SDQ) | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  The Strengths and Difficulties Questionnaire (SDQ) is used to assess mental health through a total difficulties score as well as through the five subscales (peer relationship problems, prosocial behavior, emotional symptoms, hyperactivity/inattention, conduct problems). The items are scored on a 3-point scale (0 to 2), and the total difficulties score is generated by summing all subscales except the prosocial scale. The summary score ranges from 0 to 40. Higher summary scores indicate more problems.
Parent: Mean change from baseline in parenting on parent-ratings of the Parenting Children and Adolescents Scale | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  The Parenting Children and Adolescent Scale has three subscales: encouragement of positive behaviors, setting limits, proactive parenting behaviors, each including 7 items. The 21 items are scored on a 5-point scale (1 to 5) and the total scale sum ranges from 21 to a maximum of 105, with a higher score indicating more positive parenting. The proactive parenting behavior-subscale at baseline is used for moderator/predictor analyses.
Parent: Mean change from baseline in parenting on parent-ratings of the Parenting Scale (over-reactivity subscale) | Pre-, mid-, and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  The Parenting Scale has one subscale that measures parental over-reactivity. The 5 items are scored on a 7-point scale (1 to 7) and the total scale sum ranges from 7 to a maximum of 35. A lower score indicates more positive parenting (after reverse coding). The Parenting Scale is included as a mediator of outcome.
Parent: Mean change in parent-ratings of family warmth | Pre-, mid-, and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  Family warmth is measured with 5 questions from the Family Check-Up Caregiver Assessment Scale. These are scored on a 5-point scale (1 to 5). Total maximum score ranges between 5 and 25. A higher score indicates a more positive relation. Warmth is included as a mediator of outcome.
Parent: Mean change in parent-ratings of family conflicts | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  Family conflicts are measured with 3 questions from the Family Check-Up Caregiver Assessment Scale. These are scored on a 7-point scale (0 to 6). Total maximum score ranges between 0 and 18. A higher score indicates larger degree of conflicts.
Parent: Mean change from baseline in parent-ratings of parental emotion regulation on the Parent Emotion Regulation Scale | Pre-, mid-, and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  Emotion regulation of the parent will be measured with the Parent Emotion Regulation Scale. The 20 items are scored on a 5-point scale (1 to 5) and are divided into four subscales: Orientation to child's emotions (5 items); Acceptance of child's and parents' emotions (4 items); Avoidance of child's emotions (6 items), Emotional lack of control (5 items). The total summary score ranges between 20 and 100 where a higher total score indicates better regulation of emotions. The subscale Emotional lack of control is included as a mediator of outcome.
Parent: Mean change from baseline in parent-ratings of child callous-unemotional traits on the Inventory of Callous-unemotional traits | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  Child callous-unemotional traits will be measured with the Inventory of Callous-unemotional traits. The 24 items are scored on a 4-point scale (0 to 3). Total sum ranges between 0-72, with higher scores indicating a greater degree of general callous-unemotional traits. The ICU has three subscales: callousness (11 items), uncaring (8 items), and unemotional (5 items).
Parent: Mean change from baseline in parent-rated child life quality on the Child Health Utility 9 Dimensions | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  Child life quality will be measured with the Child Health Utility 9 Dimensions (CHU9D).The 9 items are scored on a 5-point scale (1 to 5). Total sum ranges between 9-45, with higher scores indicating a greater degree life quality.
Parent: Mean change from baseline in parental well-being on the Depression Anxiety and Stress Scale-21 (DASS21) | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  Parents indicate their emotional negative state on the Depression Anxiety and Stress scale-21, which consists of 21 items that are rated on a 4-point scale (0 to 3). A higher total score indicates greater overall distress, with a maximum score of 63. The scale includes three subscales: Depression (0-21), Anxiety (0-21) and Stress (0-21). Scores are doubled to allow for comparison with the 42-item DASS-scale.
Child/youth: Mean change from baseline in child-ratings of child wellbeing on the Strengths and Difficulties Questionnaire (SDQ) | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program)
  Child-ratings of Strengths and Difficulties Questionnaire are used to assess mental health through a total difficulties score as well as through the five subscales (peer relationship problems, prosocial behavior, emotional symptoms, hyperactivity/inattention, conduct problems). The items are scored on a 3-point scale (0 to 2), and the total difficulties score is generated by summing all subscales except the prosocial scale. The summary score ranges from 0 to 40 where higher summary scores indicate more severe problems.
Child/youth: Mean change from baseline in child-ratings of child life quality on the Child Health Utility 9 Dimensions | Pre- and post-interventions (5 and 15 weeks after the initiation of the internet-based parent support program)
  Child life quality will be measured with the Child Health Utility 9 Dimensions (CHU9D).The 9 items are scored on a 5-point scale (1 to 5). Total sum ranges between 9-45, with higher scores indicating a greater degree life quality.
Parent: Mean change in ratings of satisfaction with the week | Weeks 0 to 15 after baseline. Completed once a week at each session.
  Three questions to parents scored 0 to 10 for those participating in an intervention, about their satisfaction with the week and with managing situations. Total maximum score ranges between 0-30, with a higher score indicating higher satisfaction.
Child: Mean change in ratings of satisfaction with the week | Weeks 6 to 15 after baseline. Completed once a week at each session.
  Three questions to children scored 0 to 10 for children participating in an intervention, about their satisfaction with the week and with how managing situations or emotions. Total maximum score ranges between 0-30, with a higher score indicating higher satisfaction.
Parental and child experiences of each session | Weeks 6 to 15 after baseline. Completed once a week at each session
  Four questions after each session about how the parent or child experienced the session and exercises. Rated on a scale 0-10, with a maximum total score ranging between 0 and 40. A higher score indicates greater satisfaction with the session.
Parent: Inventory of health-related costs | Pre- and post-intervention (15 weeks after the initiation of the internet-based parent support program), and six months after the final intervention.
  Treatment inventory of costs in patients with psychiatric disorders (Tic-P) collects information about medical costs and productivity losses, and includes questions about health care use, treatments, paid and unpaid labour. In this study it is used for parents of children with behavior problems. The scale is used for a health-economic evaluation of the stepped-care model and includes no summary scores.

OTHER OUTCOMES:
Parent: Background information | Pre-intervention
  Parents are asked for brief demographic information (e.g., parental age, education; child age, gender, attention deficit hyperactivity disorder [adhd]-diagnosis). A total of 13 questions. Child age, gender and adhd-diagnosis are used for moderator/predictor analyses.
Parent: Background information about number of limited prosocial emotions (callous-unemotional traits) | Pre-intervention
  Parents are asked about the number of child limited prosocial emotions. A total of 4 items answered yes/no (total sum between 0-4). Used for moderator/predictor analyses.
Parent: Number of participants with oppositional defiant disorder or conduct disorder diagnosis | Pre-intervention
  Oppositional defiant disorder diagnosis or Conduct disorder diagnosis (limited to presence of aggressive symptoms and serious violations of rules). This variable is used as moderator/predictor.
Use of each intervention: number of sessions, homework tasks | From pre- to post-interventions (between 6 to 15 weeks after the initiation of the intervention)
  A summary of the mean number of sessions and homework tasks completed during each intervention.
Drop-out rate | From pre- to post-intervention (6 to 15 weeks after the initiation of the intervention)
  The drop out from the interventions (number of participants)
Experiences of the interventions through individual qualitative interviews with parent and youth | After the interventions are completed, about 15-20 weeks after the initiation of the first intervention
  Qualitative interviews with 20 parents and 20 youth who want to participate after the Step 2-intervention will explore parent's and child's/youth's experiences of the stepped care model and the interventions. Satisfaction, feasibility, acceptability, and relevance of the interventions are investigated.
Parent and child: Closing questions about the intervention | Post-intervention (measured between 6 to 10 weeks after the initiation of the intervention)]
  Closing questions about satisfaction, relevance, and usefulness of the intervention. Parents and children respond to four questions rated on a scale 0-10, with a maximum total score ranging between 0 and 40. A higher score indicates greater satisfaction.
Parent: Closing question about possible negative effects of the interventions | Post-intervention (measured 15 weeks after the initiation of the internet-based intervention)
  Parents are asked whether any negative effects have been experienced from any of the interventions (scored yes/no). If yes, parents are asked to describe the negative experience, and the extent the family was affected a) during the intervention, b) today (each scored 0-3; higher scores indicating a more negative experience).
Parent: Information about participation in interventions | Post-intervention (measured 15 weeks after the initiation of the internet-based intervention)
  Parents are asked to provide information on what interventions the family has participated in during the past 10 weeks, such as courses, internet-based or group-based support, individual or group-based child support, or other interventions, and the extent of these.
Clinician: perception of implementation | Weeks 6 to 15 after baseline. Completed once a week at each session.
  Clinicians will respond to six questions rated 0-10 after each session during Step 2 about their adherence to and implementation of the manual and treatment. Higher scores indicate higher satisfaction with implementation (maximum weekly mean score is 60).

CONTACTS AND LOCATIONS:
Overall Officials: Pia Enebrink, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No